CLINICAL TRIAL: NCT06948500
Title: Effectiveness of an Immersive Virtual Reality-based Therapeutic Exercise Program With Altered Visual Feedback in Patients With Fibromyalgia: A Randomized Controlled Trial
Brief Title: Effectiveness of an IVR-based Therapeutic Exercise Program With Altered Visual Feedback in Fibromyalgia Patients
Acronym: IVR-F
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Chair Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-80; CEEI25/643 (Other: Universidad CEU Cardenal Herrera)
Record Dates: First submitted 2025-04-10; First posted 2025-04-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Immersive Virtual reality; Exercise; Pain
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality + Physical Activity (Experimental): A set of ten therapeutic exercises using IVR will be implemented. These exercises are designed to enhance strength, stability, mobility, and flexibility in the abdomino-lumbo-pelvic region and lower limbs. During each exercise, participants will wear IVR goggles that modify visual proprioceptive feedback by altering the perceived range of movement. Specifically, the visual input provided by the IVR system will create a discrepancy between actual physical movement and perceived motion, allowing participants to visually experience movements differently from reality.
  Interventions: Other: Immersive Virtual Reality; Other: Physical Activity
- Physical Activity (Active Comparator): Control-group participants will perform the same 6-week therapeutic-exercise program as the experimental group; the only difference will be the absence of the IVR. Training methodology, load progression, assessment procedures, and physiotherapist supervision will remain identical, ensuring comparability between groups.
  Interventions: Other: Physical Activity

INTERVENTIONS:
Other: Immersive Virtual Reality — Participants will wear an HTC Vive Pro head-mounted display with waist, hand and foot trackers during 60-min sessions, 2 times/week for 6 weeks (12 sessions). A gender- and skin-tone-matched first-person avatar will be calibrated to the user's anthropometrics and will mirror all real-time movements. Standardised audio instructions will be played through the headset; a virtual mirror will provide visual feedback.
  To facilitate lumbar mobility, two sensorimotor illusions will be applied: (1) Flexion illusion: Avatar upper-limb length will be reduced by ≈20%, encouraging greater trunk flexion; (2) Extension illusion: A virtual bar will rise with lumbar extension but will under-represent real movement by ≈10%. Both manipulations will update continuously throughout each repetition. A physiotherapist will supervise every session and will record adverse events.
  Arms: Immersive Virtual Reality + Physical Activity
Other: Physical Activity — Participants will undertake a 6-week therapeutic exercise program, consisting of two sessions per week (12 sessions total), with a primary objective of reducing fibromyalgia's impact on daily life. Each session will involve ten exercises performed in one or two sets each, depending on the week of the protocol. Exercise repetitions and intensity will be individualized using the Borg Rating of Perceived Exertion (RPE) scale (6-20), maintaining an intensity range of RPE 13-17. Specifically, intensity will start at RPE 14 (moderate) in Weeks 1-2, increase to RPE 15 (moderate-high) in Weeks 3-4, and peak at RPE 16 (high) in Weeks 5-6. No external load will be applied during the first three weeks to allow participants to adapt to the program, while progressive resistance will be introduced during the final three weeks according to individual capacity, ensuring a safe and gradual overload.

SUMMARY:
The primary aim of this randomized controlled trial is to determine the efficacy of a 6-week immersive virtual reality (IVR)-based therapeutic exercise intervention, which manipulates visual proprioceptive input during exercise, for patients diagnosed with fibromyalgia (FM). Participants will be randomly allocated into two groups: an experimental group performing therapeutic exercises integrated with IVR featuring modified visual feedback, and a control group executing identical exercises without IVR integration. The primary outcome will assess the impact of fibromyalgia on daily activities, while secondary outcomes will comprehensively evaluate fatigue, sleep quality, severity of fibromyalgia symptoms, health-related quality of life, anxiety and depressive symptoms, fear-avoidance beliefs, pain catastrophizing, kinesiophobia, indicators of central sensitization, lumbar spine flexion and extension range of motion, somatosensory function, body perception distortion, muscle strength of the handgrip and quadriceps, functional mobility, lower limb strength, behavioral regulation concerning exercise adherence, and patient-reported experiences regarding IVR use. This trial seeks to elucidate whether incorporating IVR into therapeutic exercise protocols reduces the impact of fibromyalgia on patients' daily lives and improves physiological, psychological, and physical outcomes compared to traditional exercise approaches without IVR.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic and multifactorial condition marked by widespread pain, fatigue, sleep disturbances, and various neurocognitive and psychosomatic symptoms, severely impacting quality of life and increasing healthcare costs. Although therapeutic exercise is a first-line, evidence-based treatment, its implementation is often hindered by low adherence, kinesiophobia, and maladaptive pain beliefs. Immersive virtual reality (IVR) has gained attention as a novel approach to enhance exercise efficacy through sensory immersion, cognitive distraction, and embodiment. Visual feedback manipulation in IVR-such as creating the illusion of reduced movement-has been shown to increase range of motion and engagement without intensifying perceived pain or effort. While non-immersive VR systems have shown benefits in symptom management and adherence, IVR appears to offer superior outcomes via real-time multisensory integration. However, no studies have yet investigated the clinical effects of integrating IVR with altered visual input during therapeutic exercise in FM. This will be a randomized controlled trial evaluating a 6-week IVR-based exercise program that modulates visual input to create the perception of reduced movement in FM patients. The experimental group will be compared to a control group following the same exercise program without IVR. Outcome measures include pain intensity, fatigue, sleep quality, kinesiophobia, functional capacity, symptom severity, and user experience. This study seeks to fill a critical gap in FM rehabilitation by testing whether IVR-enhanced exercise with visual modulation reduces the impact of fibromyalgia on patients' daily lives and improves physiological, psychological, and physical outcomes compared to traditional exercise approaches without IVR.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with fibromyalgia according to any of the classification criteria established by the American College of Rheumatology (ACR), including those from 1990, 2010, 2011, or 2016;
* Ability to communicate effectively with the research staff;
* A self-reported pain intensity score of ≥3 on a 11-point Numerical Pain Rating Scale (NRS-11).

Exclusion Criteria:

* Presence of comorbidities and/or symptoms that constitute a contraindication for immersive virtual reality or exercise-based interventions;
* Presence of medical conditions that may interfere with study outcomes, such as visual, auditory, perceptual, or sensory disorders;
* Use of medications that could potentially affect study results;
* Engagement in another therapeutic physical activity program during the intervention period, or any modifications to existing therapies (including medication or physical therapy) throughout the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact | At six weeks
  Measured with Spanish version of the Revised Fibromyalgia Impact Questionnaire (FIQR). This 21-item instrument evaluates physical function (0-30), overall impact (0-20), and symptom severity (0-50), yielding a total score from 0 to 100, with higher scores indicating greater impairment.

SECONDARY OUTCOMES:
Fatigue | At six weeks
  Fatigue will be assessed using the Spanish version of the Multidimensional Fatigue Inventory (MFI-20), a validated 20-item self-report instrument measuring five dimensions: general and physical fatigue, reduced activity and motivation, and mental fatigue. Items are scored on a 5-point Likert scale, yielding total scores from 20 to 100, with higher scores indicating greater fatigue.
Sleep quality | At six weeks
  Measured using the validated Spanish version of the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-report measure evaluating sleep over the past month across seven components. Total scores range from 0 to 21, with higher scores indicating poorer sleep.
Pain distribution | At six weeks
  Assessed with the Widespread Pain Index (WPI; 0 - 19), the 19 item body map component of the 2016 ACR Fibromyalgia criteria. Participants mark each anatomical region in which they have experienced pain during the previous week; the total score corresponds to the number of painful sites, ranging from 0 (no pain) to 19 (pain in all sites), with higher scores indicating a wider pain distribution and greater disease burden.
Symptom severity | At six weeks
  Measured with the Symptom Severity Scale (SSS; 0 - 12), the second component of the 2016 ACR Fibromyalgia criteria. Participants rate the severity of fatigue, non-restorative sleep, cognitive problems and extent of additional somatic symptoms on 0 to 3 Likert items (0 = none, 3 = severe). Scores are summed to yield a total ranging from 0 (no symptoms) to 12 (maximal severity), with higher values reflecting a greater symptom severity.
Change in Fibromyalgia Survey Diagnostic Criteria (FSDC) total score | At six weeks
  The FSDC total score will be calculated by summing the Widespread Pain Index (WPI) and Symptom Severity Scale (SSS) scores. This yields an aggregate score ranging from 0 to 31, with higher values reflecting a greater overall fibromyalgia symptom burden.
Health-related quality of life | At six weeks
  Measured using the Spanish EQ-5D-5L, a validated self-reported tool measuring five dimensions on five severity levels. Responses yield an index score (-0.5 to 1.0), with lower values indicating worse health, calculated using the Spanish value set.
Anxiety and depression | At six weeks
  Assessed using the Spanish version of the Hospital Anxiety and Depression Scale (HADS), a 14-item self-report tool comprising two subscales, HADS-Anxiety and HADS-Depression, each scored 0-21. Items are rated on a 4-point Likert scale (0-3), with higher scores indicating greater severity.
Pain catastrophizing | At six weeks
  Measured using the Spanish version of the 13-item Pain Catastrophizing Scale (PCS), which evaluates the frequency of catastrophic thoughts and feelings related to pain across three subscales: rumination, magnification, and helplessness. Items are rated from 0 to 4, yielding a total score of 0-52, where higher scores indicate greater catastrophizing.
Fear-avoidance beliefs | At six weeks
  Assessed using the Spanish version of the 16-item Fear-Avoidance Beliefs Questionnaire (FABQ), scored on a 7-point Likert scale (0-6), where higher scores indicate stronger avoidance beliefs.
Kinesiophobia | At six weeks
  Assessed using the Spanish version of the Tampa Scale for Kinesiophobia (TSK-11), an 11-item self-report measure of fear of movement and reinjury. Items are scored on a 4-point Likert scale (1-4), with total scores ranging from 11 to 44. Higher scores indicate greater kinesiophobia.
Central sensitization | At six weeks
  Measured using the Central Sensitization Inventory (CSI), a validated 25-item self-report measure assessing symptoms associated with central sensitization. Scores range from 0 to 100, with scores of 40 or higher indicating the presence of a central sensitization syndrome.
Pressure Pain Threshold | At six weeks
  Assessed with a handheld digital algometer (Force One™, Wagner Instruments). Measurements will be taken at two sites: (1) the dorsal surface of the right third finger, midway between the distal and middle interphalangeal joints; and (2) a point 5 cm lateral to the right of the spinous process of the third lumbar vertebra (L3). A 1 cm² rubber tip will apply steadily increasing force until the participant first perceives pain; the force will be recorded in kilograms (kg). Three trials will be performed at each site, with 30 seconds of rest between trials, and the mean of the three readings for each site will be used for analysis. Lower pressure pain threshold (PPT) values (kg) indicate higher pain sensitivity. Higher PPT values indicate lower pain sensitivity.
Temporal summation of pain | At six weeks
  Measured with a handheld digital algometer (Force One™, Wagner Instruments) applied to the dorsal surface of the right third finger. Ten pressure pulses, each rising at 2 kg·s-¹ to the individual's mean pressure pain threshold, will be delivered at 1 Hz. Participants will rate pain intensity on a 0-10 verbal Numeric Rating Scale after the first and tenth pulses. The temporal summation (TS) score is calculated as NRS₁₀ - NRS₁ (range: -10 to +10), with positive values indicating temporal summation of pain, a marker of central sensitization.
Conditioned pain modulation | At six weeks
  Assessed with a cuff-induced ischemic stimulus on the left upper arm. The cuff is inflated at 20 mm Hg·s-¹ until the first pain sensation, held for 30 seconds, then adjusted to maintain a pain intensity of 3/10 on the Numeric Rating Scale (NRS), and kept inflated. While the cuff remains on, a digital algometer delivers 10 pressure pulses to the dorsal surface of the right third finger: rising at 2 kg·s-¹ to the site-specific mean pressure pain threshold (PPT), held for 1 second, with 1 second of rest between pulses. Pain intensity is rated (0-10 NRS) after the first and tenth pulses. The conditioned pain modulation (CPM) effect is expressed as NRS₁₀ - NRS₁ (range -10 to +10). Lower or more negative values denote weaker endogenous pain inhibition.
Lower limb strength and endurance | At six weeks
  Assessed using the 30-Second Sit-to-Stand Test (STS-30), a functional test that evaluates lower limb strength and endurance by measuring an individual's ability to repeatedly rise from a chair without upper limb support over a 30-second period. The total number of repetitions performed during the 30-second period serves as an indicator of functional capacity, with higher scores reflecting better performance.
Functional mobility | At six weeks
  Assessed using the Timed Up and Go (TUG) Test, a widely used clinical tool that evaluates gait speed, dynamic balance, and overall functional capacity. Participants are timed while rising from a chair, walking three meters, turning around, walking back, and sitting down. Shorter times indicate better functional performance.
Isometric quadriceps strength | At six weeks
  Measured using a handheld dynamometer, a widely applied tool for quantifying neuromuscular function in individuals with fibromyalgia. The portable device will be placed just above the ankle while the participant is seated with the knee flexed at 90°, in order to measure maximal voluntary isometric contraction (MVIC) of the quadriceps muscle.
Handgrip strength | At six weeks
  Measured with a Jamar hydraulic dynamometer, according to the protocol described by Hamilton et al. Participants will sit with feet flat on the floor, shoulder adducted and neutrally rotated, elbow flexed at 90°, and wrist and forearm in a neutral position. Three maximal trials will be performed with verbal encouragement, with at least 4-minute rest intervals between attempts. The average of the three trials will be used for analysis.
Behavioral regulations in exercise | At six weeks
  Motivational regulation was assessed using the Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3), a 24-item self-report instrument grounded in Self-Determination Theory. Each item is rated on a 5-point Likert scale (0 = "not true for me" to 4 = "very true for me"), producing six subscale scores-Amotivation, External Regulation, Introjected Regulation, Identified Regulation, Integrated Regulation, and Intrinsic Regulation-each ranging from 0 to 16. The total raw score ranges from 0 to 96, with higher values reflecting stronger endorsement of the statements. Depending on the pattern of subscale scores, elevated Intrinsic and Integrated Regulation scores indicate more autonomous motivation, whereas higher External Regulation and Amotivation scores denote more controlled or amotivated regulation.
Dizziness provoked by immersive virtual-reality | At six weeks
  Dizziness will be monitored at every session using a 0-10 Numeric Rating Scale (NRS), where 0 indicates "no dizziness" and 10 indicates "worst imaginable dizziness." Dizziness will be captured as a continuous safety outcome, as it is expected to be the most frequent adverse effect of VR. Documenting its intensity will allow for timely adjustments to the intervention protocol. Higher scores will indicate greater levels of dizziness experienced during VR use.
Change in pain intensity from pre- to post-exercise session (11-point Numeric Rating Scale, 0-10) | Immediately before and after each exercise session over the 6-week intervention period (two sessions per week).
  Pain intensity will be recorded immediately before and after each exercise session using an 11-point Numeric Rating Scale (NRS-11) ranging from 0 ("no pain") to 10 ("worst imaginable pain"). Participants will be asked: "On a scale from 0 to 10, how intense is your pain right now?". Higher scores indicate greater pain intensity. The outcome will be calculated as the within-session change in pain (post-exercise minus pre-exercise score).
Change in total physical activity (MET-minutes/week) | At six weeks
  Total weekly physical activity will be estimated using the International Physical Activity Questionnaire - Short Form (IPAQ-SF), a 7-item self-report tool validated in Spanish and recommended by the World Health Organization. Participants report the frequency and duration of walking, moderate, and vigorous physical activities over the previous seven days. Minutes of walking are weighted by 3.3 METs, moderate activity by 4.0 METs, and vigorous activity by 8.0 METs. These values are summed to yield a total MET-minutes-per-week score. The possible range is from 0 to no upper limit; higher values indicate greater energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Lisón, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Juan Fco. Lisón, Valencia, Valencia-valència, Spain